CLINICAL TRIAL: NCT03494010
Title: Hybrid Closed-Loop Insulin Delivery System in Type 1 Diabetes Candidates for a Living Donor Kidney Transplant
Status: Withdrawn | Type: Observational
Why Stopped: PI was unable to enroll anyone.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000022558
Record Dates: First submitted 2018-03-23; First posted 2018-04-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes, Type 1
Keywords: Kidney Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- prospective cohort: Patients will be followed to determine the impact of the hybrid closed-loop (HCL) system that was prescribed at part of clinical care.
  Interventions: Other: Observation
- historical controls: Medical record data of these patients, who did not use the HCL system, will be compared with patients in the HCL cohort.

INTERVENTIONS:
Other: Observation — There is no intervention. Patients will receive the HCL system as part of their clinical care.
  Groups: prospective cohort

SUMMARY:
The investigators' primary aim is to determine the impact of using hybrid closed-loop (HCL) system in patients with type 1 diabetes (T1D) and end stage renal disease (ESRD) prior to kidney transplantation.

The investigators will also determine whether HCL, by improving glucose control, will affect short-term (1 month) and long-term (12 months) complications after kidney transplantation in patients with T1D.

DETAILED DESCRIPTION:
The investigators plan to recruit up to 25 patients with type 1 diabetes (T1D) being evaluated for a living donor kidney transplantation. These patients will be followed up to 1 year after the surgery. Participants will be recruited from the Yale Transplantation Center. Patients with end stage renal disease (ESRD) and T1D referred to the pre-transplantation clinic who have a living kidney donor and who are being considered candidates for a hybrid closed-loop (HCL) system as part of routine care, will be asked to participate in this study. Patients who show interest in the HCL system are already being referred to the Yale Transplant-Endocrine Clinic and/or the Yale Diabetes Center to be evaluated for feasibility of using the HCL. Patients will also be approached about the study, once prescribed the HCL 670G system, to be used until the surgery, as standard of care (SOC).

The HCL system will be prescribed as part of a standard care for patients with T1D willing to optimize their glucose control prior to surgery. The HCL system will not be provided by the research investigators. Also as part of SOC, Medtronic® will provide initial training (1st month) and technical support for the patients. Plan for routine care use: The HCL system will be removed during the hospital admission for the transplantation surgery and restarted after hospital discharge. Participants will be followed at the Yale Diabetes Center (YDC) and/or the Yale Transplant-Endocrine Clinic (YTEC) for management of diabetes and management of HCL system.

Patients will be seen monthly prior to the kidney transplantation. After the surgery, they will come to the YDC/YTEC clinics monthly for the first 3 months and every 3 months afterwards.

Patient information to be collected as part of the study:

1. Demographics
2. Blood glucose control test results: hemoglobin A1c, fasting glucose levels
3. Other blood and urine test results pertinent to the protocol, such as: complete blood count (CBC), chemistry, kidney and liver function tests, glomerular filtration rate (GFR), urinary protein/albumin
4. HCL system and continuous glucose monitoring (CGM) report: average glucose, standard deviation (SD), indices of glucose variability (coefficient of variation), in target glucose levels, auto-mode, frequency of hypo and hyperglycemia, insulin dose and duration of use
5. Hospitalizations: peri- and post-op hyperglycemia, hypoglycemia, infections, graft rejection, other complications/morbidity, length of stay, readmissions, mortality

The results from this cohort of patients with T1D treated with the HCL undergoing kidney transplantation will be compared to a retrospective cohort of up to 25 patients. This control cohort will be identified through a Joint Data Analytics Team (JDAT) query of patients followed at the Yale Transplant Center aged between 18-65 year, with T1D and who had received a living donor kidney transplantation in the last 3 years prior to the start date of this protocol. Medical records from these patients will be reviewed by the PI and/or co-investigators. Pertinent demographic and medical information will be recorded, as described above for the HCL treated group.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Recipient of (historical controls) or on waiting list for (cohort) a living donor kidney transplant.

Exclusion Criteria:

* Cohort and Historical Controls:

  * Vision, hearing impairment (patients cannot recognize the pump and sensor signals and alarms)
  * Cognitive impairment (unless 24-hour caregiver is available)
  * Total daily insulin dose requirements less than 8 units per day
  * Patients who are not willing to check their blood glucose test at least twice a day
  * Not followed/do not plan be followed at Yale New Haven Hospital
* Cohort:

  * No living donor candidate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes who have had (historical controls) or who plan to have (cohort) a living donor kidney transplant at Yale New haven Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Duration of use of hybrid closed-loop (HCL) system | up to 1 year post-surgery
  Use will be measured in weeks

SECONDARY OUTCOMES:
Kidney transplantation outcome - graft rejection | Up to 3 months post-transplant
Kidney transplantation outcome - infections | Up to 3 months post-transplant
Kidney transplantation outcome - mortality | 3 years from study enrollment
hyperglycemia: glucose levels > 180 milligrams per deciliter (mg/dL) | change from baseline to 1 month after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
hyperglycemia: glucose levels > 180 mg/dL | change from baseline to 1 year after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
hypoglycemia: glucose levels <70 mg/dL | change from baseline to 1 month after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
hypoglycemia: glucose levels <70 mg/dL | change from baseline to 1 year after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
hemoglobin A1c | change from baseline to 1 month after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
hemoglobin A1c | change from baseline to 1 year after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
fasting glucose levels | change from baseline to 1 month after surgery
  Blood samples taken from study subjects will be used to measure this outcome.
fasting glucose levels | change from baseline to 1 year after surgery
  Blood samples taken from study subjects will be used to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Belfort De Aguiar, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Organ Transplant Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No